CLINICAL TRIAL: NCT02000973
Title: Effects of Thoracic Epidural Anesthesia With Different Local Anesthetics on Propofol Induction
Brief Title: Effects of Epidural Local Anesthetics on Propofol Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Jun Wang, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20131012
Record Dates: First submitted 2013-11-22; First posted 2013-12-04 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: General Anesthesia; Propofol Target-controlled Infusion; Thoracic Epidural Anesthesia
MeSH Terms: interventions — Lidocaine; Bupivacaine; Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal saline (Placebo Comparator): General anesthesia combined with thoracic epidural 0.9% normal saline 8ml
  Interventions: Drug: Normal Saline
- Lidocaine (Experimental): General anesthesia combined with thoracic epidural 1% lidocaine 8ml
  Interventions: Drug: Lidocaine
- Bupivacaine (Experimental): General anesthesia combined with thoracic epidural 0.25% bupivacaine 8ml
  Interventions: Drug: Bupivacaine
- Ropivacaine (Experimental): General anesthesia combined with thoracic epidural 0.3% ropivacaine 8ml
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Lidocaine — General anesthesia combined with thoracic epidural 1% lidocaine
  Arms: Lidocaine
Drug: Bupivacaine — General anesthesia combined with thoracic epidural 0.25% bupivacaine
  Arms: Bupivacaine
Drug: Ropivacaine — General anesthesia combined with thoracic epidural 0.3% ropivacaine
  Arms: Ropivacaine
Drug: Normal Saline — General anesthesia combined with thoracic epidural 0.9% normal saline
  Arms: Normal saline

SUMMARY:
The investigators designed a prospective, randomized, placebo-controlled study to determine whether thoracic epidural anesthesia(TEA) with different local anesthetics has different influences on the propofol dose during induction.

ELIGIBILITY:
Inclusion Criteria:

Surgery for thoracotomies, BMI: 18-25 Kg/m2, American Society of Anesthesiologists(ASA) classification I or II.

Exclusion Criteria:

liver or kidney disease, alcohol dependence, take sedative recently, contraindications for epidural anesthesia.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Study Chair — Dept. of Anesthesiology, First Hospital of China Medical University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (6) | 57 (6) | 57 (6) | 58 (6) | 56 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 8 | 35
  Male | 10 | 12 | 11 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Propofol Effect-site Concentration
Description: The effect-site concentration of propofol when loss of consciousness during propofol target-controlled infusing(TCI) induction of anesthesia.
Time Frame: Before starting anesthesia to finishing endotracheal intubation
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Number analyzed (Participants) | 20 | 20 | 20 | 20
ug/ml | 1.76 (0.44) | 1.14 (0.35) | 1.09 (0.39) | 1.04 (0.18)

2. Secondary Outcome: Mean Arterial Pressure
Description: The mean arterial pressure of each patient was recorded at five different time points
Time Frame: Before starting anesthesia to finishing endotracheal intubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmHg
  Baseline | 96.40 (13.82) | 99.65 (12.41) | 98.95 (11.92) | 98.25 (13.14)
  20minites after epidural injection | 99.55 (14.65) | 96.25 (10.95) | 95.90 (10.95) | 95.40 (1.94)
  Loss of consciousness | 86.75 (16.68) | 81.15 (7.53) | 81.05 (9.19) | 80.95 (12.87)
  Before endotracheal intubation | 67.15 (12.87) | 62.30 (12.05) | 61.65 (8.72) | 60.60 (7.97)
  After endotracheal intubation | 96.82 (17.57) | 84.68 (16.25) | 85.82 (10.63) | 86.12 (12.83)

3. Secondary Outcome: Heart Rate
Description: The heart rate of each patient was recorded at five different time points
Time Frame: Before starting anesthesia to finishing endotracheal intubation
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Number analyzed (Participants) | 20 | 20 | 20 | 20
beats per minute
  Baseline | 71.70 (9.53) | 69.65 (8.66) | 69.00 (8.71) | 74.80 (13.60)
  20 minites after epidural injection | 73.95 (10.94) | 69.15 (7.81) | 67.40 (8.91) | 71.50 (11.88)
  Loss of consciousness | 69.90 (8.67) | 70.40 (11.13) | 65.90 (7.25) | 70.00 (9.35)
  Before endotracheal intubation | 64.15 (9.33) | 61.75 (12.93) | 59.10 (7.63) | 61.85 (8.54)
  After endotracheal intubation | 88.00 (12.59) | 76.70 (14.24) | 75.10 (10.67) | 79.45 (10.99)

4. Secondary Outcome: Bispectral Index Score
Description: The bispectral index(BIS) score of each patient was recorded at two different time points. BIS values varies from 0 to 100(0, no cerebral activity; 40 to 60, general anesthesia; 60 to 85, sedated; 85 to 100, awake).
Time Frame: Before starting anesthesia to finishing endotracheal intubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale
  Baseline | 96.67 (1.63) | 96.70 (1.49) | 97.07 (1.41) | 96.94 (1.18)
  20 minutes after epidural injection | 96.20 (2.34) | 90.00 (6.33) | 92.43 (4.47) | 89.12 (5.61)

ADVERSE EVENTS:
Time Frame: Before starting anesthesia to finishing endotracheal intubation
Arm/Group | Normal Saline | Lidocaine | Bupivacaine | Ropivacaine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes